CLINICAL TRIAL: NCT06399757
Title: A Phase 1/2 Study to Assess the Safety and Antitumor Activity of APL-5125 in Adults With Selected Advanced Solid Tumors
Brief Title: A Study to Investigate APL-5125 in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Apollo Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP10CP01
Record Dates: First submitted 2024-05-01; First posted 2024-05-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer; Cholangiocarcinoma; Appendiceal Adenocarcinoma; Pancreatic Adenocarcinoma; Gastric Adenocarcinoma; Endometrial Adenocarcinoma; Triple Negative Breast Cancer; Ovarian Cancer; Prostate Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Cholangiocarcinoma; Adenocarcinoma, Mucinous; Triple Negative Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase 1: Dose Escalation (Experimental): Dose escalation with increasing dose levels of APL-5125 to identify Recommended Phase 2 Dose.
  Possibility to expand into select populations
  Interventions: Drug: APL-5125
- Phase 2: Dose Expansion/Optimization (Experimental): At least 2 dose levels of APL-5125 in a selected population
  Interventions: Drug: APL-5125

INTERVENTIONS:
Drug: APL-5125 — APL-5125 is an oral drug (capsule) taken daily in 28-day cycles

SUMMARY:
This is an open-label, Phase 1/2 study to determine the safety, tolerability, and efficacy of APL-5125 for the treatment of selected locally advanced or metastatic solid tumors with particular focus on Colorectal carcinoma (CRC).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Phase 1: Histologically confirmed locally advanced, inoperable, or metastatic tumor; Colorectal carcinoma, Cholangiocarcinoma, Appendiceal adenocarcinoma.
* For Phase 1 sub-studies: Colorectal carcinoma, Cholangiocarcinoma, Appendiceal adenocarcinoma, Pancreatic Adenocarcinoma, Gastric Adenocarcinoma, Endometrial Adenocarcinoma, Triple Negative Breast Cancer, Ovarian Cancer, Prostate Cancer
* Phase 2: Colorectal carcinoma
* No available standard of care therapy or participant is ineligible for standard of care therapy, except in CRC tumor type in which participant must have previously received all the following therapeutic agents:

  * fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy
  * an anti-VEGF therapy
  * if wt-RAS (wt-KRAS and wt-NRAS), an anti-EGFR therapy
* Eastern Cooperative Oncology Group (ECOG) ≤1
* Body Weight ≥40 kg.
* Female participants of childbearing potential must have negative serum pregnancy test at screening; must not plan to become pregnant or have ova harvested or breastfeed while on study; must be willing to use specific contraception or avoid intercourse
* Male participants must be willing to use specific contraception and not plan to impregnate a female partner or donate sperm while on study
* Participant must be willing and able to provide written informed consent and to comply with the requirements of the trial

Exclusion Criteria:

* Certain medical conditions such as: active brain metastases, carcinomatous meningitis, unstable angina pectoris, myocardial infarction or clinically significant ventricular arrhythmias, symptomatic congestive heart failure, uncontrolled active infection, history of significant hemorrhage within 4 weeks of the first dose date, intestinal disease or major gastric surgery, arterial thrombosis within 6 months of screening
* Certain prior therapies such as: anti-cancer treatment within 2 weeks of Cycle 1 Day 1, prior radiotherapy within 14 days before screening, active anti-coagulation therapy, over the counter or prescription medications within 14 days or 5 half-lives prior to cycle 1 day 1, herbal medicines and supplements within 14 days
* Major surgery within 1 month of screening
* Hemoglobin < 9.0 g/dL
* Absolute neutrophil count < 1.5 x 10^9/L
* Platelet count < 100 x 10^9/L
* Hepatic function:

  1. Aspartate aminotransferase and/or alanine aminotransferase (ALT) >3 × upper limit of normal (ULN) (>5 x ULN for subjects with liver metastases)
  2. Total bilirubin >1.5 × ULN (except participants with Gilbert's syndrome).
  3. Albumin < 3 g/dL
* Calculated or measured creatinine clearance of <60 mL/minute calculated using the formula of Cockcroft and Gault ([140 - Age] × Mass [kg] / [72 × serum creatinine mg/dL]). Multiply result by 0.85 if female.
* Fridericia's corrected QT interval (QTcF) >470 msec or a family history of Long QT Syndrome.
* Cardiac function: Echocardiogram (or MUGA) showing Left Ventricular Ejection Fraction (LVEF) <45% at rest
* Infectious diseases: positive for HIV (unless controlled with active retroviral therapy), hepatitis B and hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Emergent Adverse Events [Safety] | Through study completion, approximately one year
  Evaluation of safety parameters including treatment emergent adverse events as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, electrocardiogram results.
Incidence of dose limiting toxicities [Tolerability] (Phase 1) | Cycle 1 Day 1 to Cycle 2 Day 1 (a cycle is 28 days)
  Evaluation of tolerability parameters including dose limiting toxicities as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs and electrocardiogram results
Determine Recommended Phase 2 Dose (RP2D) levels of APL-5125 in participants with selected advanced solid tumors (Phase 1) | Approximately one year
Assess the anti-tumor activity of APL-5125 in patients with Colorectal carcinoma (Phase 2) | Response is assessed every 8 weeks; after one year of treatment, response is assessed every 12 weeks. (Assessed for up to 2 years.)
  Response is assessed per RECIST version 1.1 criteria

SECONDARY OUTCOMES:
Assess the preliminary anti-tumor activity of APL-5125 in colorectal carcinoma patients (Phase 1) | Response is assessed every 8 weeks; after one year of treatment, response is assessed every 12 weeks. (Assessed for up to 2 years.)
  Response is assessed per RECIST version 1.1 criteria
Assess the pharmacokinetics (PK) of APL-5125 (Phase 1) | On days 1, 2, 4, 8, 15 of cycle 1, and on day 1 of cycle 2 and cycle 3 (a cycle is 28 days).
  Evaluate PK parameters: oral clearance
Assess the pharmacokinetics (PK) of APL-5125 (Phase 1) | On days 1, 2 ,4, 8, 15 of cycle 1, and on day 1 of cycle 2 and cycle 3 (a cycle is 28 days).
  Evaluate PK parameters: volume of distribution
Evaluate biomarker(s) in the tumor | Through study completion, approximately one year
  Assessment of biomarker(s) in pre- and post-treatment tumor tissue
Further assess the anti-tumor activity of APL-5125 (Phase 2) | Response is assessed every 8 weeks; after one year of treatment, response is assessed every 12 weeks. (Assessed for up to 2 years.)
  Response is assessed per RECIST version 1.1 criteria
Incidence of treatment emergent adverse events [Further Safety] (Phase 2) | Through study completion (approximately 2 years)
  Evaluation of safety parameters including treatment emergent adverse events as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, electrocardiogram results
Further assess the PK of APL-5125 (Phase 2) | On days 1 and 8 of cycle 1, and on day 1 of cycle 2 and cycle 3 (a cycle is 28 days).
  Evaluate PK parameters: oral clearance
Further assess the PK of APL-5125 (Phase 2) | On days 1 and 8 of cycle 1, and on day 1 of cycle 2 and cycle 3 (a cycle is 28 days).
  Evaluate PK parameters: volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Aggarwal, MD, Study Chair — Apollo Therapeutics Ltd
Locations (9):
- United States (9):
  - City of Hope, Duarte, California
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Florida Cancer Specialists & Research Institute, Sarasota, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Duke Cancer Institute, Durham, North Carolina
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas
  - NEXT Oncology- San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No